CLINICAL TRIAL: NCT06262659
Title: Effect Of Blood Flow, Vascular Diameter, And Depth Measurements With Intraoperative Doppler Ultrasonography On Arteriovenous Fistula Maturation In Dialysis Patients: A Prospective Study
Brief Title: The Effect of Ultrasonography on Blood Flow,Vessel Diameter,and Depth Measurements in Dialysis Patients With Fistula
Status: Completed | Type: Observational
Sponsor: Kudret Atakan Tekin (Other)
Responsible Party: Sponsor-Investigator, Kudret Atakan Tekin, Principal Investigator, Hitit University
Organization: Hitit University (Other)
Other Study IDs: 2023-142
Record Dates: First submitted 2024-02-05; First posted 2024-02-16 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Arteriovenous Fistula
Keywords: arteriovenous fistula; fistula flow; vascular diameter; intraoperative Doppler Ultrasound; arteriovenous fistula maturation
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group fistula: Preoperative age, gender, weight, height, body mass index, diabetes mellitus, hypertension, asthma, smoking status, postoperative chest pain, intraoperative AVF flow, AVF depth, AVF vascular diameter, and postoperative 6th-week Doppler ultrasonography measurements of AVF flow, AVF depth, and AVF vascular diameter will be recorded for the patients included in the study. Maturation assessment will be made based on these results.
  AVF flow measurement will be performed intraoperatively and at the 6th week postoperatively using Doppler ultrasonography (B-Mode and duplex ultrasound on the LOQIC; GE Healthcare Technologies, Milwaukee, Wisconsin, United States). For each patient, AVF flows will be recorded by taking at least 3 measurements of AVF flow, depth, and vascular diameters at 2, 5, 10, and 15 cm proximal to the AVF anastomosis, and arithmetic averages will be calculated.
  Interventions: Other: Doppler Ultrasonography Assessment

INTERVENTIONS:
Other: Doppler Ultrasonography Assessment — Preoperative data will be collected from the latest available data within the last month. Preoperative Doppler ultrasonography venous mapping for all patients will be performed by experienced Radiology Specialists.
  AVF flow measurement will be performed intraoperatively and at the 6th week postoperatively using Doppler ultrasonography (B-Mode and duplex ultrasound on the LOQIC; GE Healthcare Technologies, Milwaukee, Wisconsin, United States). For each patient, AVF flows will be recorded by taking at least 3 measurements of AVF flow, depth, and vascular diameters at 2, 5, 10, and 15 cm proximal to the AVF anastomosis, and arithmetic averages will be calculated. AVF flow will be expressed in "ml/min," and the vascular structure diameters and the distance of AVF from the skin will be indicated in "mm." AVF depth will be calculated as the distance from the skin to the anterior wall of the AVF.

SUMMARY:
Arteriovenous fistulas (AVF) are considered essential and the primary vascular access for end-stage renal disease patients to receive hemodialysis (HD) treatment. The maturation failure rate of AVFs is approximately 23%. The aim of our study is to compare intraoperative fistula flow and measurements of vascular structures' diameters with postoperative fistula maturation, following the completion of the fistula operation, to reveal the relationship between them. Providing insights into the need for intraoperative intervention and/or postoperative fistula management based on these measurements is intended to contribute to the literature by offering predictions and perspectives.

DETAILED DESCRIPTION:
Arteriovenous fistulas (AVF) are generally acknowledged as the 'gold standard' for hemodialysis (HD) access in end-stage renal disease patients. While they exhibit the most successful performance, their lifespan is longer compared to other access types, and the infection and hospitalization rates are lower. However, it is known that many newly created fistulas do not mature to a level that provides sufficient HD access. There is no universal definition for a matured AVF, and the method adopted in the updated National Kidney Foundation's Kidney Disease Outcomes Quality Initiative (NKF-KDOQI) guidelines is widely used. KDOQI has defined the "6s rule" to describe maturation (a flow rate of 600 ml/min, an AVF located within 6 millimeters from the skin surface to facilitate successful and repeatable cannulation by HD staff, and finally, a minimum diameter of 6 millimeters). A matured AVF should be continuously cannulated and allow a minimum blood flow of 300-400 ml per minute. Various patient factors, including Diabetes Mellitus (DM), female gender, and age, have been suggested to be associated with poor AVF maturation. However, these factors are less important when preoperative ultrasound mapping of the relevant arterial and venous region shows vessels of sufficient size. Preoperative ultrasound venous mapping has been proven to significantly assist in deciding on an AVF with a higher chance of successful maturation. Surgical or endovascular intervention is frequently required for AVFs that do not mature or to facilitate maturation. Even after successful AVF maturation, interventions are often needed to maintain long-term patency in hemodialysis. The maturation of AVF typically takes between 6 to 8 weeks. Previous studies have evaluated postoperative ultrasound criteria to assess AVF maturation and determine the need for interventions that would promote maturation. These studies reported high predictive values for AVF maturation using postoperative blood flow thresholds of 420-800 ml/min or diameters of 3.6-5.4 mm. However, the generalizability of these studies is limited due to the relatively small number of patients, the prevalence of radiocephalic AVFs, and variable definitions of AVF maturation. While published studies have focused on the value of postoperative AVF ultrasound measurements in predicting maturation, none have assessed the predictive value for determining primary patency (the time until the first intervention when the AVF achieves independent maturation). Venous diameter maturity is an independent determinant, and a venous diameter less than 2.5 mm is often associated with non-maturation, especially if the vein cannot expand after tourniquet application; a preoperative ultrasound measurement of a vein ≥4 mm is expected to result in successful maturation. A series of 158 patients reported that venous diameter was the main independent determinant of functional maturation, and it was the only independent variable. NKF-KDOQI guidelines suggest allowing a fistula to mature for at least one month before cannulation. Cannulating within 14 days after AVF creation reduces long-term fistula survival and increases the risk of subsequent fistula failure by 2.1 times compared to fistulas cannulated after 14 days. Fistulas cannulated between 15 and 28 days showed no significant difference in non-maturation rates compared to those cannulated after 43 to 84 days. Ultrasound is a non-invasive imaging technology that can significantly contribute to understanding vascular anatomy in the context of dialysis access. Depth measurements and flow volume detections in arterial flow, in particular, can guide interventions. Postoperative ultrasound is commonly used to assess AVF maturation for hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of AVF for hemodialysis due to end-stage renal failure,
* Patients aged 18 and older but younger than 70,
* Patients who have not undergone dialysis before,
* Patients with normal sinus rhythm on EKG,
* Patients with triphasic flow in upper extremity arterial Doppler ultrasonography,
* Patients with a minimum vessel diameter of ≥2 mm for arteries and ≥2.5 mm for veins on Doppler ultrasonography.

Exclusion Criteria:

* Patients with reduced ejection fraction (EF) (<50%),
* Patients with heart valve disease,
* Patients with coronary artery disease or those who have undergone coronary artery bypass grafting surgery,
* Patients with a history of fistula creation,
* Patients undergoing fistula revision,
* Patients with peripheral vascular disease,
* Patients with venous embolism/thrombosis or occlusion history in the upper extremity superficial/deep venous system, superior vena cava,
* Patients with arterial embolism or occlusion in the upper extremity,
* Patients with burn scars in the upper extremity,
* Patients with atrophy/paralysis/plegia in the upper extremity,
* Patients with uncontrolled diabetes,
* Patients with connective tissue disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing the first-time autologous arteriovenous fistula creation surgery in end-stage renal failure will be included in the study.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
intraoperative Arteriovenous Fistula Flow Measurement | 1 hour
  AVF flow measurement will be conducted intraoperatively using Doppler ultrasonography (B-Mode and duplex ultrasound on the LOQIC; GE Healthcare Technologies, Milwaukee, Wisconsin, United States). For each patient, AVF flows will be recorded by taking at least 3 measurements of AVF flow, at 2, 5, 10, and 15 cm proximal to the AVF anastomosis, and arithmetic averages will be calculated. AVF flow will be expressed in "ml/min".

CONTACTS AND LOCATIONS:
Locations (1):
- Kudret Atakan Tekin, Merkez, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No